CLINICAL TRIAL: NCT02405650
Title: Visceral Adiposity and Physical Fitness in CKD
Brief Title: CRIC-Visceral Adiposity and Physical Fitness in Chronic Kidney Disease
Acronym: CRIC-VAP
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Pennsylvania (Other); Case Western Reserve University (Other); University of Michigan (Other); University of Illinois at Chicago (Other); University of Maryland (Other); MetroHealth Medical Center (Other); The Cleveland Clinic (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Sankar Navaneethan, PI, Baylor College of Medicine
Other Study IDs: 37396 CRIC VAP
Record Dates: First submitted 2015-03-25; First posted 2015-04-01 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Renal Insufficiency, Chronic; Obesity
Keywords: CKD, chronic kidney disease, CRIC
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum, blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRIC VAP cohort: If eligible, the participant will have additional testing at regular annual CRIC Visit. The following will occur:
  * abdominal and pelvic Magnetic Resonance Imaging (MRI) scan
  * 400 meter walk test for physical fitness

SUMMARY:
Obesity and chronic kidney disease (CKD) are major public health problems. In contrary to observations in general population, higher body mass index in those with pre-existing CKD is associated with lower mortality. Chronic Renal Insufficiency Cohort (CRIC) is an ongoing observational study to examine the consequences of CKD with a particular focus on cardiovascular illness like myocardial infarction (heart attack) and stroke. Among CRIC study participants, the investigators propose to obtain visceral and subcutaneous adiposity and physical fitness measures and study its associations with patient-centered outcomes. This study will help the investigators understand the independent and combined effects of visceral adiposity and physical fitness on cardiovascular disease, renal disease progression and death among those with CKD. Further, it will identify mechanisms that could be targeted to reduce the detrimental effects of visceral adiposity in those with kidney disease.

DETAILED DESCRIPTION:
Obesity and chronic kidney disease (CKD) are major public health problems. Obesity independent of its relationship with diabetes and hypertension is associated with the development and progression of kidney disease. However, higher body mass index (BMI) in those with pre-existing CKD is associated with lower mortality (obesity paradox). This may be due to the inability of BMI to differentiate fat mass and muscle mass, which may have opposite relationship with cardiovascular disease and death. Body fat distribution is a major factor of metabolic health with metabolic abnormalities correlating better with visceral than subcutaneous adipose tissue. Further, higher fitness levels among those with higher BMI is associated with a lower prevalence of cardiovascular risk factors and mortality that might explain this obesity paradox. Therefore, among Chronic Renal Insufficiency Cohort (CRIC) study participants, the investigators propose (a) to examine whether visceral adiposity is associated with a higher incidence of composite outcomes (i.e., mortality, cardiovascular events, end stage renal disease, and 50% decline in estimated glomerular filtration rate), (b) to determine if physical fitness modifies the association between adiposity and outcomes, and (c) to study whether visceral adiposity and physical fitness are associated with altered adipokine profile, inflammation, insulin resistance, and oxidative stress. The study proposes to enroll 526 patients with varying degrees of kidney disease from 7 clinical centers involved in the CRIC study. Visceral adiposity will be measured by magnetic resonance imaging (MRI) of the abdomen using a standard protocol, and physical fitness will be measured using a 400 m walk test during routine CRIC study visits. Results from this study will help the Investigators understand the independent and combined effects of visceral adiposity and physical fitness on cardiovascular disease and kidney disease progression among CKD patients. This study will also highlight potential pathways that mediate the relationship between adiposity and outcomes, which will become the focus of future therapeutic investigations in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-79
* Estimated Glomerular Filtration Rate 20-74 ml/min/1.73m^2

Exclusion Criteria:

* Pacemaker
* Metallic prosthesis or foreign body (joints, heart valves, clips)

  *Sites may include patients with cardiac stents and/or dental implants based on the local Radiology department criteria i.e. if there are no restrictions, they can include patients with stents and/or dental implants. If the Radiology department mandates the type of stent details and/or dental implants, site coordinator should provide this to the local Radiology department and obtain permission before enrolling the subject.
* Severe claustrophobia
* Severe osteoarthritis (use of walker or other assisted devices)

  *Sites may include patients with cane (single or quad).
* Recent cardiovascular or cerebrovascular events (within 6 months prior to enrollment)
* Kidney transplant
* Currently on dialysis
* Peripheral vascular disease limiting long distance walking

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must be participant in Prospective Cohort Study of Chronic Renal Insufficiency (CRIC). CRIC participants are a racially and ethnically diverse group of adult patients with mild-to-moderate CRI.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2015-04; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Composite of mortality, cardiovascular events, End Stage Renal Disease (ESRD) and 50% decline in estimated glomerular filtration rate (eGFR) | 5 years
  Since visceral adiposity is related to both cardiovascular disease and kidney function and to adequately power the study, we chose the composite end-point.

SECONDARY OUTCOMES:
All-cause death | 5 years
  Death details are obtained from linkage of the CRIC study with the National Death Index.
Cardiovascular events (acute myocardial infarction, congestive heart failure, cardiac arrhythmias, peripheral vascular disease and cerebrovascular events) | end of the study
  Once a patient reports a clinical event or hospitalization during the study visit, de-identified charts are adjudicated by review of hospital records by two physician reviewers and linkage with other national database
Renal events - End Stage Renal Disease plus 50% decline in Glomerular filtration rate (GFR) | 5 years
  Incident End Stage Renal Disease is being defined as initiation of chronic dialysis or kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sankar Navaneethan, M.D., Principal Investigator — Baylor College of Medicine
Locations (10):
- United States (10):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins University - ProHealth, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Case Western Reserve University, Cleveland, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Scientific & Data Coordinating Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas